CLINICAL TRIAL: NCT07334717
Title: An Observational Clinical Study to Collect Photographic Data of Wounds With Hypergranulation to Aid Development of a Hypergranulation Clinical Endpoint and Assessment Tool, And Generate Participant Reported Data to Inform Trial Design
Status: Recruiting | Type: Observational
Sponsor: Ennogen Healthcare Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: EHCI HG 04-01; 365713 (Other: Integrated Research Application System)
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Wound Complications
Keywords: Hypergranulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wounds that will be studied include venous leg ulcers, burns and complex surgical wounds.
  Interventions: Diagnostic Test: Hypergranulation Tool Proforma; Device: Device to take 2D images of wounds to allow for construction of a 3D image of the wound to assess degree of hypergranulation

INTERVENTIONS:
Diagnostic Test: Hypergranulation Tool Proforma — This is an observational study, no IMP will be used. Patients will continue to receive best evidenced based care.
  Patients will attend clinic 2-4 times. Investigators will use the Hypergranulation Tool Proforma as designed by a roundtable of clinical experts at each clinic visit to clinically assess wounds for the degree of hypergranulation present. The wound will be clinically reviewed based on 5 parameters. This enables clinicans to quantify the degree of hypergranuation of wounds and allow for assessment of wound healing over clinic visits. This will be compared to 3D images of the wound and already validated Patient Reported Outcome Forms (PROMIS) will be competed and exit patient interviews.
  The data collected will aim to validate a method for assessment of hypergranulation of wounds in the clinical setting to help inform future Phase II clinical trials.
Device: Device to take 2D images of wounds to allow for construction of a 3D image of the wound to assess degree of hypergranulation — This is an observational study, no IMP will be used. Patients will continue to receive best evidenced based care. Patients will attend clinic 2-4 times. Images using a device creating 2D images to allow for a 3D image to be created of the wound. The 3D image will allow for assessment of the volume/ height of hypergranulation and the percentage of the wound affected. This will also produce data on the use of 3D in assessing wound healing over the clinic visits.
  investigators will also use the Hypergranulation Tool Proforma as described above and the already validated Patient Reported Outcome Forms (PROMIS) will be competed and exit patient interviews. The data collected will aim to validate a method for assessment of hypergranulation of wounds in the clinical setting to help inform future Phase II clinical trials.

SUMMARY:
Hypergranulation (HG) is well documented and a known barrier to wound healing. Accurate clinical assessment of wounds is crucial in managing HG and evaluating treatment response. Currently there is no standardised assessment for healthcare professionals to assess the severity of HG. Through a modified Delphi process involving wound care clinical experts, a prototype Hypergranulation Tool has been developed to be used in clinical practice. The Hypergranulation Tool allows assessors to grade HG within wounds as mild, moderate and severe, based on 5 separate parameters. A prospective multi-site observational study based in the United Kingdom of 80-100 adult and paediatric patients with HG within venous leg ulcers (VLU) or complex surgical wounds (CSW) will allow performance testing of the Hypergranulation Tool. Study nurses will assess wounds with the Hypergranulation Tool across 2-4 clinic visits. Data from the use of the tool will be compared with quantitative 3D analysis of the wounds, patient reported outcome and patient interview data, to help determine the validity of the Hypergranulation Tool in the clinical setting. Results from the Observational Study will inform design changes to the Hyergranulation Tool as well as the design of future HG intervention trials.

ELIGIBILITY:
Inclusion Criteria

* Male or female participants between 2 to 85 years of age (both inclusive).
* Willing and able to provide written informed consent or assent (as applicable) as evidenced by signature on the participant's consent/assent form. In case if the child is providing assent, a caregiver or LAR must sign an informed consent.
* A chronic HG wound which can be:

  * a VLU unhealed for a minimum of 6 weeks, but no longer than 24 weeks
  * an unhealed surgical wound that has been unhealed for at least 2 weeks but no longer than 24 weeks
  * a device entering the skin (eg, gastrostomy, suprapubic catheter, tracheostomy etc) that exhibits HG.
* A degree of HG that is estimated to be raised at least 2 mm above the natural skin level, or above the base of the wound and an area of HG extending at least 10 mm in its longest length.
* For VLU and surgical wounds, the wound should not have been healed by at least 25% area or length.
* Have good general health as defined by:

  * medically fit enough to complete the study assessments
  * free of any other systemic condition that in the opinion of the Study Investigator may have an impact on the safety of the participant.
* Be willing and able to attend all scheduled clinical assessments, (adults or caregiver)
* able to communicate well with the Study Investigator and willing and able to comply with the expectations of the study.

  * This includes gastrostomy; suprapubic catheters, tracheostomy, other tube/catheter skin entry or exit sites, abdominal surgical wound, pilonidal sinus surgical site, split-skin donor site, plastic surgery sites, healing burn sites, peri-anal surgical wounds, gastrointestinal stoma, other.

Exclusion Criteria

* Unable to provide informed consent or assent
* Unable to complete the scheduled study treatments and assessments
* Have been previously recruited into this study
* Participants who are < 2 years or >85 years of age

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 80-100 participants who meet the inclusion criteria will be be recruited into the study. Participants will be recruited from tissue viability clinics, burns clinics and wound care clinics across the North West of England.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To determine the performance of 3-D photographs as a tool to assess HG wound tissue as compared to Hypergranulation Tool Proforma clinical asssesment | August 2026
  3D images will be compared to the clinical assessment by the Hypergranulation Tool Proforma which assesses wounds based on 5 components (bleeding and friability, colour, height, exudate, and size [percentage of wound affected])

SECONDARY OUTCOMES:
To conduct and evaluate the assessment of wound healing percentage through 3-D photography compared to Study Investigator assessment with the Hypergranulation Tool | August 2026
To determine the performance of 3-D photographs in assessing HG wound tissue coverage compared to assessments made by a Study Investigator with the Hypergranulation Tool Proforma | August 2026
To assess the participant reported experience of HG of wound tissue through participant reported outcomes (PROs) and participant interviews | August 2026
To determine the performance of 3-D photographs in assessing height of HG wound tissue compared to assessments made by a Study Investigator with the Hypergranulation Tool | August 2026
To assess study-emergent adverse events (AEs) that are linked to study assessments. | August 2026

CONTACTS AND LOCATIONS:
Locations (1):
- EMS Healthcare, Ellesmere Port, Cheshire, United Kingdom